CLINICAL TRIAL: NCT02353793
Title: Trauma Patients and Hypothermia in the Emergency Room: a Trial Between Self-warming ReadyHeat® Blanket and Traditional Cotton Wool Blanket
Brief Title: Trauma Patients and Hypothermia in the Emergency Room: ReadyHeat® Versus Cotton Wool Blanket
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Timo Iden, M.D., University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ReadyHeat
Record Dates: First submitted 2014-12-15; First posted 2015-02-03 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Hypothermia; Trauma
Keywords: Hypothermia; (Poly) Trauma; Emergency Room; Warming Blanket
MeSH Terms: conditions — Hypothermia; Wounds and Injuries; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReadyHeat® blanket (Experimental): Patient warming with ReadyHeat® blanket
  Interventions: Device: ReadyHeat® blanket
- Cotton wool blanket (Active Comparator): Patient warming with cotton wool blanket
  Interventions: Device: Cotton wool blanket

INTERVENTIONS:
Device: ReadyHeat® blanket — Using ReadyHeat® blanket for patient warming
  Arms: ReadyHeat® blanket
Device: Cotton wool blanket — Using cotton wool blanket for patient warming
  Arms: Cotton wool blanket

SUMMARY:
Hypothermia is a common problem in traumatized patients leading to severe complications such as impaired coagulation, increased rate of wound infections and overall patient discomfort among others. Therefore, the investigators test out the new self warming ReadyHeat® blanket device against the currently used cotton wool blanket in terms of effects on the prevention and treatment of hypothermia.

DETAILED DESCRIPTION:
Hypothermia is a common problem in traumatized patients leading to severe complications such as impaired coagulation, increased rate of wound infections and overall patient discomfort among others. Therefore, the investigators test out the new self warming (via an exothermic reaction) ReadyHeat® blanket device against the currently used cotton wool blanket in terms of effects on the prevention and treatment of hypothermia. Near body core temperature is measured by a sublingual sensor as the "gold standard" of body core temperature measurement - the pulmonary artery catheter - is too invasive and not suited for this collective of patients in the emergency room setting. Blanket use will be randomized. Temperature will be taken at emergency room admission, after 15, 30 and 45 minutes of treatment as well as right before handing the patient over to the next caring unit (ICU, IMC, operating theatre etc.). If treatment time is shorter than expected measurement will stop at the latest possible point. Blankets will be applied to the patient once admission in the emergency room is complete and will only be lifted for interventions.

ELIGIBILITY:
Inclusion Criteria:

- Trauma patients ≥ 18 years of all severity stages including poly traumatized patients admissioned through the emergency room

Exclusion Criteria:

* Patients < 18 years
* Patients after pre-hospital cardiac arrest or ongoing CPR at time of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Body core temperature at the end of completed emergency room treatment | When handing the patient over to the next caring unit (ICU, operating theatre etc.) n most cases an average time frame < 60 min is maintained
  Body core temperature taken after completed emergency room treatment incl. imaging. In most cases an average time frame < 60 min is maintained.

SECONDARY OUTCOMES:
Body core temperature during emergency room treatment | Temperature measurement: Admission, after 15, 30, 45 minutes
  Body core temperature taken after emergency room admission and 15, 30 and 45 minutes after beginning of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jan Höcker, M.D., Study Director — Klinik für Anästhesiologie und Operative Intensivmedizin, Arnold-Heller-Str. 3, Haus 12, 24105 Kiel
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Curry N, Davis PW. What's new in resuscitation strategies for the patient with multiple trauma? Injury. 2012 Jul;43(7):1021-8. doi: 10.1016/j.injury.2012.03.014. Epub 2012 Apr 7. PMID 22487163
- [Background] Sessler DI. Temperature monitoring and perioperative thermoregulation. Anesthesiology. 2008 Aug;109(2):318-38. doi: 10.1097/ALN.0b013e31817f6d76. PMID 18648241
- [Background] Kapan M, Onder A, Oguz A, Taskesen F, Aliosmanoglu I, Gul M, Tacyildiz I. The effective risk factors on mortality in patients undergoing damage control surgery. Eur Rev Med Pharmacol Sci. 2013 Jun;17(12):1681-7. PMID 23832738